CLINICAL TRIAL: NCT06541379
Title: Investigation of the Effect of Motor Imagery Ability on Upper Extremity Functionality and Proprioception in Transradial Amputees Using Myoelectric Prostheses
Brief Title: Effect of Motor Imagery Ability on Functionality and Proprioception in Amputees Using Myoelectric Prostheses"
Status: Recruiting | Type: Observational
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Ayse Yazgan, Lecturer, Medipol University
Other Study IDs: MedipolU-OP-AY-01
Record Dates: First submitted 2024-08-01; First posted 2024-08-07 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Amputation of Upper Limb Below Elbow; Prosthesis User
Keywords: Imagery; Amputee; Prosthetic; Functional; Myoelectric

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Transradial Amputees Using Myoelectric Prosthesis: The Standardized Mini Mental Test (SMMT) will be used to assess the cognitive status of individuals, the Beck Depression Inventory (BDI) to assess depression symptoms, the Movement Imagery Questionnaire-3 to assess motor imagery ability, the Mental Chronometry Test (MKT) to measure motor imagery time, the mobile application called "Orientate" to assess hand mental rotation task performance, the Box and Block Test to assess gross motor dexterity and functionality, the Jebsen Taylor Hand Function Test (JTEFT) to assess fine and gross motor functions of the hand, the Disabilities of the Arm Shoulder and Hand (DASH) for upper extremity functional assessment, the Modified Functional Reach Test (MFUT) to measure the dynamic balance of the trunk and the Joint Position Sense measurement to assess proprioceptive sense.
  Interventions: Other: No intervention
- Control Healthy Group: The Standardized Mini Mental Test (SMMT) will be used to assess the cognitive status of individuals, the Beck Depression Inventory (BDI) to assess depression symptoms, the Movement Imagery Questionnaire-3 to assess motor imagery ability, the Mental Chronometry Test (MKT) to measure motor imagery time, the mobile application called "Orientate" to assess hand mental rotation task performance, the Box and Block Test to assess gross motor dexterity and functionality, the Jebsen Taylor Hand Function Test (JTEFT) to assess fine and gross motor functions of the hand, the Disabilities of the Arm Shoulder and Hand (DASH) for upper extremity functional assessment, the Modified Functional Reach Test (MFUT) to measure the dynamic balance of the trunk and the Joint Position Sense measurement to assess proprioceptive sense.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention

SUMMARY:
The purpose of this study is to evaluate the motor imagery ability in transradial amputees using myoelectric prosthesis, compare it with the control group and investigate its effect on functionality and proprioception.

DETAILED DESCRIPTION:
In the sensory and motor homunculus, the upper extremity, especially the hand, areas cover a larger area. Morphological changes occur in the body in amputees due to upper extremity amputation. In addition, neural restructuring occurs due to the lack of sensory input and visual feedback. These neurophysiological changes experienced in amputees affect the cortical areas of the brain. This situation can also negatively affect motor imagery ability. For this reason, upper extremity prosthesis systems with different control mechanisms have been developed. In one of the developed systems, myoelectric prostheses, since the signals received with electrodes due to muscle contraction provide sensory input to amputees, known that it increases synaptic sprouting in the brain and improves motor imagery ability. There are studies that use motor imagery in stroke, spinal cord injury, Parkinson's disease, postoperative anterior cruciate ligament injuries, cervical and lumbar region pain problems. In addition, it focused on motor imagery after amputation and emphasized that the evidence on whether motor imagery ability is impaired in amputees is not sufficient. In a study, it was found that the use of upper extremity prosthesis increases the hand mental rotation ability and this situation is related to the body integrity of amputees with the use of prosthesis. After investigatorsexamination and screening, to the best of investigators knowledge, no study was found that evaluated the motor imagery ability of transradial amputees using myoelectric controlled prosthesis and examined its effect on functionality. Therefore, the aim of investigators study is to evaluate the motor imagery ability in transradial amputees using myoelectric prosthesis, compare it with the control group and investigate its effect on functionality and proprioception. Transradial amputees using myoelectric prosthesis and the control group (healthy individuals) between the ages of 22-65 will be included in the study. Demographic information of all participants to be included in the study will be recorded with the "Case Assessment Form". Standardized Mini Mental Test (SMMT) to evaluate the cognitive status of individuals, Beck Depression Inventory (BDI) to evaluate depression symptoms, Movement Imagery Questionnaire-3 to evaluate motor imagery ability, Mental Chronometry Test (MKT) measuring motor imagery time, "Orientate" mobile application to evaluate hand mental rotation task performance, Box and Block Test to evaluate gross motor hand skills and functionality, Jebsen Taylor Hand Function Test (JTEFT) to measure upper extremity functions,Disabilities of the Arm Shoulder and Hand (DASH) for upper extremity functional assessment, Modified Functional Reach Test (MFUT) to measure dynamic balance of the trunk, and Joint Position Sense measurement to evaluate proprioceptive sense will be used. All data will be evaluated by statistical analysis methods.

ELIGIBILITY:
Inclusion Criteria:

Amputee group inclusion criteria

* Being an amputee using a unilateral transradial and myoelectric prosthesis
* Having at least 6 months of prosthesis experience
* Having a maximum score of 15 on the Beck Depression Inventory
* Having a minimum score of 26 on the Standardized Mini Mental Test
* Being willing to participate in the study

Control Group inclusion criteria

* Being between the ages of 18-65
* Having a minimum score of 26 on the Standardized Mini Mental Test
* Having signed the Informed Voluntary Consent Form
* Having a maximum score of 15 on the Beck Depression Inventory
* Being literate

Exclusion Criteria:

Amputee group exclusion criteria

* Having another physical problem other than amputation
* Having a diagnosed cognitive disorder
* Not being able to read or write

Exclusion criteria for the control group from the study

* Having any neurological, orthopedic, psychological (such as schizophrenia, psychosis) and systemic problems
* Having an unchangeable visual or auditory disability

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Being an amputee using a unilateral transradial and myoelectric prosthesis and control group
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Movement Imagination Questionnaire-3 | immediately after screening
  In order to determine the imagery ability of all individuals included in the amputee and control groups, the "Movement Imagery Questionnaire-3" developed and validated and validated in Turkish will be used (internal consistency coefficient: 0.87). With the 12 items in this questionnaire, internal visual imagery, external visual imagery and kinesthetic imagery abilities will be assessed through four actions each. The actions will be actively performed by the individuals at the beginning. Then, they were asked to perform these actions as mental tasks. These mental tasks were scored using a seven-point Likert scale (1: very difficult to see, feel; 7: very easy to see, feel). In the calculation of the score, the average score of the four relevant actions will be taken for each of the three sub-dimensions.

SECONDARY OUTCOMES:
Orientate Mobile Application | immediately after screening
  It is used for the purpose of evaluating mental rotation. It is based on the principle of showing individuals hand images from different angles with the application. There are a total of 25 hand images for the test. Participants will be asked to sit comfortably in a chair in front of a table and the mobile application will be opened and the test will be applied. Participants will be asked to decide which of the images is the right and which is the left hand photo as soon as possible. At the end of the test, the application will show the number of correct answers, the number of incorrect answers, the number of missed answers and the time to complete the test. The accuracy rates will also be recorded by comparing the number of correct answers to the total number of images.
Box and Block Test | immediately after screening
  The box and block test is a method used to evaluate gross motor skills and measure functionality. For the test, 150 blocks with dimensions of 2.5 cm and a box divided into two compartments are used. Participants will be asked to take the blocks one by one from the box consisting of two compartments on a table and see how many blocks they can put into the empty compartment placed in the other compartment in 60 seconds, and the results will be noted. In order for the evaluation to be accurate, the process will be repeated three times and the average of the recorded evaluation will be taken.
Jebsen Taylor Hand Function Test (JTEFT) | immediately after screening
  It is a performance-based test developed in 1969 that includes movements in daily life activities. It includes different types of grip and evaluates the speed of individuals in these tasks. The materials for the test are standardized and can be easily accessed in the clinic. Participants will be asked to do 7 different tasks in the test content. These tasks are writing, turning cards, picking up objects, eating, stacking checkers, picking up light wide objects and picking up heavy wide objects. Participants will be asked to do each task separately with both hands. The test score will be calculated by recording the time it takes for participants to complete the tasks.
Modified Functional Reach Test (MFUT) | immediately after screening
  It is a test developed to evaluate the dynamic balance and functionality of the trunk. The distance the trunk can extend forward and sideways without losing balance in a sitting position is measured. The participants will be measured next to a wall with participants ankles, knees, and hips at 90° flexion and participants feet in full contact with the ground. In the relevant position, the arm will be extended parallel to the wall, then extended forward and sideways, and the distance in between will be recorded in cm with the help of a tape measure.
Disabilities of the Arm Shoulder and Hand (DASH) | immediately after screening
  It is a scale that measures the activity and participation limitations of the upper extremity. It is based on the principle of self-assessment of the results. In 2006, the validity and reliability study of the survey in Turkish was conducted. There are 11 questions in the survey. It aims to question the difficulties that individuals have during participants daily living activities. The answers are scored from good to bad on a Likert scale, with each answer being scored from 1 to 5. The survey has options such as 1 = no difficulty, 2 = mild difficulty, 3 = moderate difficulty, 4 = extreme difficulty, and 5 = unable to do at all.
Joint Position Sense Measurement | immediately after screening
  Joint position sense is evaluated with the aim of measuring the ability of a certain joint angle to be repeated in an individual. This measurement can be applied passively-actively or with eyes closed-open. This test reveals the acuity of defining a certain angle in joints. Considering the amputation level of transradial amputees included in investigators study, shoulder and elbow joint position sense of all participants will be measured.
Mental Chronometry Test | immediately after screening
  It is known as another method that can be used to evaluate motor imagery ability. Mental chronometry is based on the principle of comparing the time it takes to perform a movement with the time it takes to mentally image the same movement. This test provides more objective results than survey applications. The Mental Chronometry test will be evaluated in investigators study with the help of the Box and Block Test. Participants will be asked to imagine this task after performing the box block test performance. The time required to collect 15 blocks will be recorded, unlike the normal procedure of the box block test. Purpose is evaluate mental chronometry ability rather than gross manual dexterity.

OTHER OUTCOMES:
Beck Depression Inventory | immediately after screening
  It is a special test designed to protect the level of the person and is available internationally. The Turkish validity and reliability study of the operation was carried out in 1988. The test consists of twenty-one items. Each maddening has 4 options as 0, 1, 2, 3. Participants are allowed to accumulate one point for all items. The total maximum score is 63. It is stated that the increase in the total score is heavy. While the score between 0-9 points is normal, 10-16 points are resistant to light violence, 17-29 points are resistant to moderate violence and 30-63 points are resistant to severe violence. People who earn a maximum of 15 points are included in investigators study.
Standardized Mini Mental Test (SMMT) | immediately after screening
  It is an assessment scale used to obtain information about the individual's individual functioning status. It was first published in 1997. It consists of thirty questions calculated out of 30 points. It is a test that evaluates cognitive status by measuring cognitive functions such as attention-gathering ability, recall, orientation, calculation, speaking, comprehension, reading, writing, memory, and drawing skills. SMMT will be added to the assessment process as an inclusion criterion, not as an outcome measure in investigators study. The highest score that can be obtained from the scale in total is 30 points. People with a score of 26 and above are considered to have normal cognitive levels.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe Yazgan, Study Director — https://www.medipol.edu.tr/
Locations (1):
- Istanbul Medipol University, Istanbul, Beykoz, Turkey (Türkiye)

REFERENCES:
- [Result] Saimpont A, Malouin F, Durand A, Mercier C, di Rienzo F, Saruco E, Collet C, Guillot A, Jackson PL. The effects of body position and actual execution on motor imagery of locomotor tasks in people with a lower-limb amputation. Sci Rep. 2021 Jul 2;11(1):13788. doi: 10.1038/s41598-021-93240-6. PMID 34215827
- See also: Reference Article Link — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC8253815/